CLINICAL TRIAL: NCT06163300
Title: MRI Analysis and Degenerative Spine
Status: Recruiting | Type: Observational
Sponsor: Universidade Nova de Lisboa (Other)
Responsible Party: Sponsor
Other Study IDs: a319_b
Record Dates: First submitted 2023-11-30; First posted 2023-12-08 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Spine Disease
MeSH Terms: conditions — Spinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Healthy volunteers
  Interventions: Diagnostic Test: MRI advanced techniques
- Disease: Patients affected by disease
  Interventions: Diagnostic Test: MRI advanced techniques

INTERVENTIONS:
Diagnostic Test: MRI advanced techniques — Participants will be submitted to MRI studies at diagnosis, during disease evolution and after treatment. Data collected will be analysed by two different neuroradiologists using advanced techniques.

SUMMARY:
Analysis of MRI advanced techniques in degenerative spinal disease.

The main questions it aims to answer are:

* Can we assess microstructural integrity of compressed nerve roots in degenerative spinal disease
* What are the image biomarkers affected by disease
* How they evolve with disease progression and treatment

ELIGIBILITY:
Inclusion Criteria:

* Age between 50 and 85 years
* Diagnosis of spinal disease by clinical and imagiological criteria
* More than 3 months duration of disease
* Ability to give consent
* Fluent portuguese speaker

Exclusion Criteria:

* Previous spine surgery
* Spinal instability
* Neurological disease that might interfere with walking
* Known orthopedic conditions that causes significant gait impairment
* Dementia or development disorder with cognitive impairment
* Inability to give consent

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with suspected diagnosis of the spinal disease in study and that meet the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
ODI - Oswestry Disability Index | 18 months
  Measured using the ODI scale (range 0 - 50)
Lumbar Pain Intensity | 18 months
  Measured using the Numeric Pain Rating Scale (range: 0 - 10 )

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital da Luz Setúbal, Setúbal, Portugal

IPD SHARING:
Plan to Share IPD: Undecided